CLINICAL TRIAL: NCT05845866
Title: Randomized Controlled Pilot Trial Targeting Weight and Shape Concern Among Women Enrolled in Behavioral Weight Management
Brief Title: Targeting Weight and Shape Concern Among Women with High Body Weight
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23DK124578 (NIH)
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Body Image Disturbance; Overweight and Obesity; Weight Loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified Body Project (Experimental): Participants will receive this four week intervention followed by 6 months of behavioral weight management
  Interventions: Behavioral: Modified Body Project; Behavioral: Lifestyle intervention for weight loss
- Facts about obesity, myths about weight loss (Active Comparator): Participants will receive this four week intervention followed by 6 months of behavioral weight management
  Interventions: Behavioral: Facts about obesity, myths about weight loss; Behavioral: Lifestyle intervention for weight loss

INTERVENTIONS:
Behavioral: Modified Body Project — The Body Project, an evidence-based body image intervention developed for young women at risk for eating pathology, was adapted for use among adult women with high weight and shape concern and high body weight who want to lose weight.
  Arms: Modified Body Project
Behavioral: Facts about obesity, myths about weight loss — This intervention is designed to help individuals prepare for weight loss and is focused on facts about obesity, myths about weight loss, and the importance of a varied diet.
  Arms: Facts about obesity, myths about weight loss
Behavioral: Lifestyle intervention for weight loss — This 24-week behavioral weight management program is based on the Look AHEAD and Diabetes Prevention Program manuals. It is designed to facilitate 7-10% weight loss of initial body weight through dietary and physical activity changes with use of behavioral strategies to support lifestyle changes over time.

SUMMARY:
This study is a randomized controlled trial to evaluate the effect of an adapted version of the Body Project program among adult women of higher body weight who want to lose weight. The study will evaluate treatment effects on weight and shape concern and explore the impact of intervention on weight loss outcomes.

DETAILED DESCRIPTION:
The objective of this study is to conduct a randomized controlled pilot trial to test the effects of a 28-week treatment protocol that combines a modified body image intervention (The Body Project: weeks 1-4) with a 6-month standard behavioral weight management treatment (weeks 5-28). The combined protocol will be evaluated in comparison to a control group that receives an education only program during weeks 1-4 followed by the same 6-month weight management treatment. It will be tested among women with high body weight who report High Weight and Shape Concern and would like to lose weight.

The goals of the study are:

1. To evaluate effects of a manualized intervention on Weight and Shape Concern prior to starting weight management.
2. To evaluate the effects of the modified Body Project intervention on momentary weight/shape-related thoughts and overeating episodes during behavioral weight management.
3. To conduct exploratory analyses comparing effects of the two treatment conditions on weight loss and other weight-related behaviors (e.g., exercise, adherence to self-monitoring).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Body Mass Index between 25-40
* Eating Disorder Examination-Questionnaire weight concern subscale greater than or equal to 4
* Eating Disorder Examination-Questionnaire shape concern subscale greater than or equal to 4.25
* Personal use of cell phone
* Able to engage in moderate intensity activity
* Desire for weight loss

Exclusion Criteria:

* No eating disorder history
* Not pregnant
* Not breastfeeding
* No childbirth/delivery within 9 months
* No substance use disorder
* No weight loss medication or history of bariatric surgery
* No other weight loss program participation

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Weight and shape concern | week 4
  Assessed using the weight concern and shape concern subscales of the Eating Disorder Examination-Questionnaire. Subscale scores range from 0-6.

SECONDARY OUTCOMES:
Momentary Weight and Shape Concern | week 16, week 28
  Ecological momentary assessment will be used to assess in-the-moment thoughts about weight and shape on a 0-10 scale.
Overeating | week 16, week 28
  Ecological momentary assessment will be used to assess overeating in daily life.

OTHER OUTCOMES:
Weight change | week 4 to week 28
  Percent weight change will be calculated from weight at the start of weight loss treatment to program completion.
Adherence to lifestyle intervention | week 4 to week 28
  Adherence to exercise, dietary tracking, and self-weighing will be monitored throughout weight loss treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States